CLINICAL TRIAL: NCT04113759
Title: Postoperative Blood Flow Restriction Training Following Hip Arthroscopy: A Randomized Clinical Trial
Brief Title: Blood Flow Restriction Following Hip Arthroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19093005
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Labral Tear, Glenoid; Femoral Acetabular Impingement
MeSH Terms: conditions — Rotator Cuff Injuries; Femoracetabular Impingement

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): The control group will receive sham BFR, in which a non-occlusive pressure is applied with the cuff. The exercises performed will be identical to the BFR group.
  Interventions: Behavioral: Sham BFR Rehabilitative Therapy
- BFR Postoperative Rehabilitation (Experimental): The experimental group will receive BFR postoperative rehabilitation, which will involve performing a series of blood flow restriction exercises identical to the control group.
  Interventions: Behavioral: Blood Flow Restriction Rehabilitative Therapy

INTERVENTIONS:
Behavioral: Blood Flow Restriction Rehabilitative Therapy — BFR cuffs placed at the proximal thigh, just inferior to the greater trochanter.
  Inflation time not to exceed 20 minutes. One BFR session per treatment. BFR exercise dosage: 4 sets of the following repetitions 30, 15, 15, 15, 30 second rest between sets, 1 min rest between exercises.
  Progress exercise if pain <2/10 on VAS and RPE <5 on 0-10 scale. (Heerey et al), and no break down in form.
  Arms: BFR Postoperative Rehabilitation
Behavioral: Sham BFR Rehabilitative Therapy — The schedule, type of exercises, repetition ranges, and other physical therapy interventions will be the same as the BFR experimental group - however a non-occlusive pressure will be applied with the cuff in the control group.
  Arms: Control Group

SUMMARY:
This study will be a prospective randomized, double-blinded, placebo-controlled trial of patients undergoing primary hip arthroscopy for FAIS and/or labral pathology. All patients who sign the consent form will be enrolled in the study and randomized to one of the two treatment arms. Follow-up will take place at 1-month, 3-months, 6-months, and 1-year.

DETAILED DESCRIPTION:
The investigators propose using standardized strength testing, serial quadriceps measurements, and MRI to assess the efficacy of BFR training in increasing muscle hypertrophy following hip arthroscopy. Investigators will perform a randomized double-blinded placebo-controlled controlled trial of patients undergoing primary hip arthroscopy. Quadriceps strength will be measured with dynamometers at 3, 6, and 12 month time points, with Biodex strength testing at 6 and 12 months, postoperatively. Additionally, standardized circumferential leg measurements to assess quadriceps hypertrophy will be performed at 1, 3, 6 and 12-month time points. Patients will also undergo a hip MRI at 6 months postoperatively to quantify muscle size and appearance about the hip joint. Patient reported outcomes including standard outcomes measures at 3, 6, and 12 months and return to work/sport data will also be collected at standard time points. Patients will also be followed longitudinally for rates of reinjury, return to work, and return to sport.

This study will evaluate the efficacy of BFR therapy in the postoperative period of primary hip arthroscopy to improve muscle hypertrophy during the short-term rehabilitation period. This will be directly measured by strength testing with dynamometers and Biodex testing. Other metrics will include standard validated patient reported outcomes at 3, 6 and 12 month time points including hip disability and osteoarthritis outcome score (HOOS), Harris Hip score (HHS), visual analog scale (VAS) for pain, international hip outcome tool (iHOT-12), and Hip outcome score (HOS), and return to sport questionnaires. Standardized serial circumferential thigh measurements will also be recorded at each visit, in additional to a one time MRI at 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-40
* English-speaking
* Clinical and radiographic examination (MRI) consistent FAIS and/or labral pathology, and are schedule for primary hip arthroscopy
* Written and informed consent for study participation

Exclusion Criteria:

* Patients younger than 18 or older than 40 years of age
* Non-native English speaker
* Revision surgery or prior history of ipsilateral hip or knee surgery
* Inability to comply with the proposed follow-up clinic visits
* Patients lacking decisional capacity
* Patients with a history of deep vein thrombosis, pulmonary embolism, or known clotting disorder or hypercoagulable state
* Pregnant or breast-feeding women. Pregnancy as determined by a positive pregnancy test prior to procedure. Females of childbearing potential must agree to use an acceptable birth control method during study participation.
* Worker's compensation patients
* Any clinically significant finding that would place the patient at health risk, impact the study, or affect the completion of the study
* Any psychiatric illness that would prevent comprehension of the details and nature of the study and interfere with follow-up clinic visits

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Quadriceps Strength | 3 month time point
  Will be measured with dynamometer
Quadriceps Strength | 6 month time point
  Will be measured with dynamometer
Quadriceps Strength | 12 month time point
  Will be measured with dynamometer
Biodex strength testing | 6 month time point
  Isokinetic strength testing
Biodex strength testing | 12 month time point
  Isokinetic strength testing
Standardized circumferential leg meaurements | 1 month time point
  To assesss quadricep hypertrophy
Standardized circumferential leg meaurements | 3 month time point
  To assesss quadricep hypertrophy
Standardized circumferential leg meaurements | 6 month time point
  To assesss quadricep hypertrophy
Standardized circumferential leg meaurements | 12 month time point
  To assesss quadricep hypertrophy
Muscle size and appearance about the hip joint | 6 months postoperatively
  To be assessed via hip MRI postoperatively

SECONDARY OUTCOMES:
Hip Disability and Osteoarthritis Outcome Score | 3 month time point
  Used to assess the patient's opinion about their hip and associated problems and to evaluate symptoms and functional limitations related to the hip during a therapeutic process.
Hip Disability and Osteoarthritis Outcome Score | 6 month time point
  Used to assess the patient's opinion about their hip and associated problems and to evaluate symptoms and functional limitations related to the hip during a therapeutic process.
Hip Disability and Osteoarthritis Outcome Score | 12 month time point
  Used to assess the patient's opinion about their hip and associated problems and to evaluate symptoms and functional limitations related to the hip during a therapeutic process.
Harris Hip Score | 3 month time point
  Gives a maximum of 100 points. Pain receives 44 points, function 47 points, range of motion 5 points, and deformity 4 points. Function is subdivided into activities of daily living (14 points) and gait (33 points). The higher the HHS, the less dysfunction.
Harris Hip Score | 6 month time point
  Gives a maximum of 100 points. Pain receives 44 points, function 47 points, range of motion 5 points, and deformity 4 points. Function is subdivided into activities of daily living (14 points) and gait (33 points). The higher the HHS, the less dysfunction.
Harris Hip Score | 12 month time point
  Gives a maximum of 100 points. Pain receives 44 points, function 47 points, range of motion 5 points, and deformity 4 points. Function is subdivided into activities of daily living (14 points) and gait (33 points). The higher the HHS, the less dysfunction.
Visual Analog Scale for pain | 3 month time point
  A 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable."
Visual Analog Scale for pain | 6 month time point
  A 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable."
Visual Analog Scale for pain | 12 month time point
  A 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable."
International hip outcome tool | 3 month time point
  Comprised of 33 questions relating to:
  Symptoms and Functional Limitations Sports and Recreational Activities Job-Related Concerns Social, Emotional, and Lifestyle Concerns
International hip outcome tool | 6 month time point
  Comprised of 33 questions relating to:
  Symptoms and Functional Limitations Sports and Recreational Activities Job-Related Concerns Social, Emotional, and Lifestyle Concerns
International hip outcome tool | 12 month time point
  Comprised of 33 questions relating to:
  Symptoms and Functional Limitations Sports and Recreational Activities Job-Related Concerns Social, Emotional, and Lifestyle Concerns
Hip Outcome Score | 3 month time point
  A self-administered questionnaire with a scoring system composed of 2 sub-scales. The Activities of Daily Living (ADL) sub-scale made of 19 items and a Sports sub-scale composed of 9 items.
Hip Outcome Score | 6 month time point
  A self-administered questionnaire with a scoring system composed of 2 sub-scales. The Activities of Daily Living (ADL) sub-scale made of 19 items and a Sports sub-scale composed of 9 items.
Hip Outcome Score | 12 month time point
  A self-administered questionnaire with a scoring system composed of 2 sub-scales. The Activities of Daily Living (ADL) sub-scale made of 19 items and a Sports sub-scale composed of 9 items.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Chahla, MD PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States